CLINICAL TRIAL: NCT00104364
Title: An Open-label, Dose Escalation Phase I/II Trial of a KSP Inhibitor Given as a Constant 24-Hour Infusion in Patients With Advanced Solid Tumors
Brief Title: A Study of MK0731 in Patients With Advanced Solid Tumors (0731-002)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0731-002; 2005_004
Record Dates: First submitted 2005-02-25; First posted 2005-02-28 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — 4-(2,5-difluorophenyl)-N-(3-fluoro-1-methylpiperidin-4-yl)-2-(hydroxymethyl)-N-methyl-2-phenyl-2,5-dihydro-1H-pyrrole-1-carboxamide

INTERVENTIONS:
Drug: MK0731

SUMMARY:
The purpose of this trial is to study MK0731 in patients with recurrent or non-responsive solid tumors, or cancers for which standard therapy does not exist.

This is an early phase trial and some specific protocol information is proprietary and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years of age with recurrent or non-responsive solid tumors, or cancers for whom standard therapy does not exist. Part of the study includes only patients who have taxane-resistant cancers.

Exclusion Criteria:

* Patients who have had treatment with any investigational therapy within the past 30 days.
* Patients who have certain types of blood cancers such as leukemia or lymphoma.
* Patients who have uncontrolled congestive heart failure (CHF), chest pains, or had a heart attack within the past 3 months, or have undergone bone marrow or stem cell transplantation.
* Patient is pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-05; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of MK0731 administered as a 24-hour CIV Infusion. Dose limiting toxicities. Maximum tolerated dose and recommended Phase II dose of L-001154704 administered as a 24 hour CIV infusion.

SECONDARY OUTCOMES:
Predose predictive biomarkers of response to MK0731

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Holen K, DiPaola R, Liu G, Tan AR, Wilding G, Hsu K, Agrawal N, Chen C, Xue L, Rosenberg E, Stein M. A phase I trial of MK-0731, a kinesin spindle protein (KSP) inhibitor, in patients with solid tumors. Invest New Drugs. 2012 Jun;30(3):1088-95. doi: 10.1007/s10637-011-9653-1. Epub 2011 Mar 22. PMID 21424701